CLINICAL TRIAL: NCT03954041
Title: A Multicenter, Double-Blind, Multidose, Placebo-Controlled, Randomized, Parallel-Group, Phase 2 Study to Evaluate the Efficacy and Safety of Intravenous BIIB093 for Patients With Brain Contusion
Brief Title: A Study to Evaluate the Efficacy and Safety of BIIB093 in Participants With Brain Contusion
Acronym: ASTRAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early completed due to strategic considerations, not for efficacy or safety reasons.
Sponsor: Remedy Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 252BN201; 2018-003858-24 (EudraCT Number)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Brain Contusion
MeSH Terms: conditions — Brain Contusion | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB093 3 mg (Experimental): Participants will be administered BIIB093 3 milligrams per day (mg/day) as a IV bolus followed by rapid and slow intravenous (IV) infusions for 96 hours.
  Interventions: Drug: BIIB093
- BIIB093 5 mg (Experimental): Participants will be administered BIIB093 5 mg/day as a IV bolus followed by rapid and slow IV infusions for 96 hours.
  Interventions: Drug: BIIB093
- Placebo (Placebo Comparator): Participants will be administered BIIB093 matching placebo as a IV bolus followed by rapid and slow IV infusions for 96 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB093 — Administered as specified in the treatment arm.
  Other Names: Glibenclamide; CIRARA; RP 1127
  Arms: BIIB093 3 mg; BIIB093 5 mg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective is to determine if BIIB093 reduces brain contusion expansion by Hour 96 when compared to placebo.

The secondary objectives are to evaluate the effects of BIIB093 on acute neurologic status, functional outcomes, and treatment requirements, to further differentiate the mechanism of action of BIIB093 on contusion expansion by examining differential effects on hematoma and edema expansion, and to determine if BIIB093 improves survival at Day 90 when compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of brain contusion with lesions within the supratentorial brain parenchyma totaling >3 mL in volume per Investigator assessment of baseline non-contrast computed tomography scan (NCCT) at Screening.
* A score of 5 to 15 on the Glasgow Coma Scale (GCS).
* Functionally independent, in the opinion of the Investigator, prior to index head injury.

Key Exclusion Criteria:

* In the judgment of the Investigator, participant is likely to have supportive care withdrawn within 24 hours.
* Indication for immediate evacuation of IPH or DC.
* Clinical signs of brainstem herniation, in the opinion of the Investigator.
* NCCT or magnetic resonance imaging (MRI) evidence of penetrating brain parenchyma. Cerebrospinal fluid leak in isolation is not exclusionary unless evidence of parenchymal penetration by an external force (e.g., blunt object, bullet, or depressed skull fracture).
* Any presence of midbrain or posterior fossa injury as assessed by imaging and clinical examination.
* Presence of concomitant spinal cord injury as assessed by imaging and clinical examination.
* Life-threatening or nonsurvivable polytrauma, per Investigator's judgment.
* Use of novel oral anticoagulants (NOACS; including direct thrombin inhibitors such as dabigatran, or Factor Xa inhibitors such as rivaroxaban or apixaban), in preceding 3 days prior to the injury, if known.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-10-06 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Remedy Pharmaceuticals
Locations (63):
- United States (25):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Scottsdale Healthcare Hospitals d/b/a HonorHealth, Scottsdale, Arizona
  - University of Arizona Medical Center, Tucson, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Medical Group Neurosurgery, Marietta, Georgia
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Northwell Health, Manhattan, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, East Providence, Rhode Island
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- France (6):
  - CHU de Brest - Hôpital de la Cavale Blanche, Brest, Finistere
  - Hopital Caremeau, Nîmes, Gard
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - CHU Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Puy De Dome
  - CHU Amiens - Hopital Sud, Amiens, Somme
- Germany (4):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Neurologische Klinik Bad Neustadt/Saale, Bad Neustadt/Saale, Bavaria
  - Universitaetsmedizin Goettingen, Göttingen, Lower Saxony
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig
- Israel (7):
  - Rabin MC, Petah Tikva, Central District
  - Health Corporation of Galilee Medical Center, Naharya, Northern District
  - Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Rambam Health Care Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Torrette, Ancona
  - ASST Monza - Ospedale San Gerardo di Monza, Monza Brianza, Milano
  - Azienda Ospedaliero Universitaria di Parma, Pama, Parma
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Ospedale Maggiore di Novara, Novara
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
- Japan (6):
  - Kimitsu Chuo Hospital, Kisarazu-Shi, Chiba
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Nara Medical University Hospital, Kashihara-shi, Nara
  - Rinku General Medical Center, Izumisano, Osaka
  - Nippon Medical School Hospital, Bunkyō City, Tokyo-to
  - Yamaguchi University Hospital, Ube-Shi, Yamaguchi
- Spain (8):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruna
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in Israel, France, Japan, Italy, Spain, and the United States.
Pre-assignment Details: A total of 92 participants were enrolled and randomized, out of which 86 participants were dosed with BIIB093 or a matching placebo.
Groups:
- Placebo: Participants were administered with BIIB093 matching placebo as an intravenous (IV) bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
- BIIB093 3 mg/Day: Participants were administered with BIIB093 up to 3 milligrams per day (mg/day) as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
- BIIB093 5 mg/Day: Participants were administered with BIIB093 up to 5 mg/day as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
Period: Overall Study
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Started | 48 | 23 | 21
Completed | 30 | 14 | 11
Not Completed | 18 | 9 | 10
Not completed — Lost to Follow-up | 3 | 3 | 6
Not completed — Death | 4 | 0 | 1
Not completed — Death by neurologic criteria | 0 | 0 | 1
Not completed — Reason not specified | 7 | 4 | 2
Not completed — Withdrew prior to dosing | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All dosed population included all the randomized participants who received any study drug (BIIB093 or a placebo).
Groups:
- Placebo: Participants were administered with BIIB093 matching placebo as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
- BIIB093 3 mg/Day: Participants were administered with BIIB093 up to 3 mg/day as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day | Total
Number analyzed (Participants) | 44 | 21 | 21 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.18) | 55.7 (19.87) | 55.0 (21.02) | 57.4 (17.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 3 | 14
  Male | 36 | 18 | 18 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4 | 8
  Not Hispanic or Latino | 39 | 15 | 14 | 68
  Unknown or Not Reported | 3 | 4 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 1
  Race: Asian | 12 | 5 | 5 | 22
  Race: Black or African American | 1 | 0 | 0 | 1
  Race: White | 26 | 12 | 13 | 51
  Race: Not Reported | 2 | 4 | 3 | 9
  Race: Other | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Total Contusion Volume (Hematoma Plus Perihematomal Edema) at 96 Hours as Measured by Brain Imaging
Description: Total contusion volume including hematoma and perihematomal edema volumes reported in milliliters (mL) was assessed by the central imaging core laboratory on baseline non-contrast computed tomography (NCCT), 24-hour NCCT, and the 96-hour scan (Magnetic resonance imaging [MRI] and/or NCCT) and the scans obtained prior to decompressive craniectomy (DC), intraparenchymal hematoma (IPH) evacuation, or comfort measures only (CMO).
Time Frame: Baseline up to 96 hours (Day 4)
Population: mITT population=all randomized participants who received any study drug (BIIB093/placebo), had at least one final read per central review of contusion volume from NCCT/MRI scan acquired between 10 hours after study drug infusion initiation and Hour 96 visit/NSx/CMO. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis. 'Number analyzed' signifies number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 38 | 20 | 19
mL
  Baseline | 29.45 (29.688) | 21.21 (26.659) | 21.33 (26.637)
  Change From Baseline at 96 Hours: number analyzed (Participants) | 34 | 19 | 15
  Change From Baseline at 96 Hours | 18.91 (23.804) | 30.07 (29.418) | 18.78 (12.771)
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; p = 0.3752, ANCOVA — P-value was analyzed by ANCOVA model with covariates: treatment, interactive response technology (IRT) stratification factors at randomization, baseline total contusion volume based on central read, imaging modality at Hour 96 (MRI vs NCCT); LS mean difference = 4.62, 95% CI 2-sided [-5.74 to 14.98]

2. Secondary Outcome: Percentage of Participants With Glasgow Outcome Scale - Extended (GOS-E) Score at Day 180
Description: The GOS-E is a global disability scale used to assess recovery after traumatic brain injury. For this study, the 8 point ordinal scale was condensed to the following 7-categories: 1 and 2 combined: Dead and Vegetative State, 3: Lower Severe disability, 4: Upper Severe disability, 5: Lower Moderate disability, 6: Upper Moderate disability, 7 : Lower Good recovery, and 8: Upper Good Recovery. Lower scores indicate death and higher scores indicate recovery.
Time Frame: Day 180
Population: mITT population included all randomized participants who received any study drug (BIIB093/placebo), had at least one final read per central review of contusion volume from NCCT/MRI scan acquired between 10 hours after study drug infusion initiation and Hour 96 visit/NSx/CMO. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 30 | 15 | 11
Percentage of participants
  Score: 1/2 | 0 | 0 | 0
  Score: 3 | 13.3 | 13.3 | 27.3
  Score: 4 | 0 | 26.7 | 9.1
  Score: 5 | 13.3 | 6.7 | 0
  Score: 6 | 26.7 | 0 | 0
  Score: 7 | 6.7 | 13.3 | 27.3
  Score: 8 | 40.0 | 40.0 | 36.4
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.40 to 3.36]

3. Secondary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Score at Day 90
Description: The mRS measures the degree of functional independence following stroke. In this study, the 7-category ordinal mRS scale was condensed to the following 5-categories: 0/1, 2, 3, 4, 5/6 where 0 and 1 reflect no disability and near-normal functioning while 5 and 6 represent severe disability and death, respectively.
Time Frame: Day 90
Population: mITT population included all randomized participants who received any study drug (BIIB093/placebo), had at least one final read per central review of contusion volume from NCCT/MRI scan acquired between 10 hours after study drug infusion initiation and Hour 96 visit or NSx or CMO, if earlier. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 39 | 19 | 14
Percentage of participants
  Score: 0/1 | 38.5 | 31.6 | 57.1
  Score: 2 | 25.6 | 26.3 | 7.1
  Score: 3 | 12.8 | 21.1 | 0
  Score: 4 | 10.3 | 15.8 | 21.4
  Score: 5/6 | 12.8 | 5.3 | 14.3
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; p = 0.4306, Regression, Logistic — P-value was analyzed by ordinal logistic regression on mRS adjusting for covariates: treatment, IRT stratification factors at randomization, baseline mRS score, and baseline total contusion volume based on central read; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.56 to 3.86]

4. Secondary Outcome: Percentage of Participants Requiring Delayed Intubation
Description: Delayed intubation is defined as participants requiring intubation (for neurologic deterioration only) at any time between 24 hours and 96 hours post-injury.
Time Frame: Day 1 (24 hours) up to Day 4 (96 hours) post-injury
Population: mITT population included all the randomized participants who received any study drug (BIIB093 or placebo) and had at least one final read per central review of contusion volume from a NCCT or MRI scan acquired between 10 hours after the initiation of study drug infusion and the Hour 96 visit or NSx or CMO, if earlier.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 44 | 21 | 20
Percentage of participants | 2.3 | 4.8 | 0

5. Secondary Outcome: Change From Baseline in Mean Total Contusion Volume (Hematoma Plus Perihematomal Edema) at 24 Hours as Measured by Brain Imaging
Description: Total contusion volume including hematoma and perihematomal edema volumes reported in mL was assessed by the central imaging core laboratory on baseline NCCT and 24-hour NCCT.
Time Frame: Baseline up to 24 hours (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 38 | 20 | 19
mL
  Baseline | 29.45 (29.688) | 21.21 (26.659) | 21.33 (26.637)
  Change From Baseline at 24 Hours: number analyzed (Participants) | 36 | 19 | 18
  Change From Baseline at 24 Hours | 8.16 (18.824) | 11.24 (13.909) | 6.67 (13.483)
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; p = 0.6478, ANCOVA — P-value was analyzed by ANCOVA model with covariates: treatment, IRT stratification factors at randomization, baseline total contusion volume based on central read; LS Mean difference = -1.53, 95% CI 2-sided [-8.19 to 5.13]

6. Secondary Outcome: Change From Baseline in Absolute Hematoma Volume at 24 Hours
Description: Hematoma volume reported in mL was assessed by the central imaging core laboratory on baseline NCCT, 24-hour NCCT, and the scans obtained prior to DC, IPH evacuation, or CMO.
Time Frame: Baseline up to 24 hours (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 40 | 20 | 20
mL
  Baseline | 6.72 (10.012) | 6.11 (12.086) | 3.62 (3.737)
  Change From Baseline at 24 Hours: number analyzed (Participants) | 38 | 19 | 19
  Change From Baseline at 24 Hours | 2.07 (5.920) | 2.13 (3.667) | 2.23 (3.537)
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; p = 0.9314, ANCOVA — P-value was analyzed by ANCOVA model with covariates: treatment, IRT stratification factors at randomization, baseline Glasgow Coma Scale (GCS) based on eCRF, and baseline absolute hematoma volume based on central read; LS Mean Difference = -0.09, 95% CI 2-sided [-2.20 to 2.02]

7. Secondary Outcome: Change From Baseline in Absolute Edema Volume at 96 Hours
Description: Edema volume reported in mL was assessed by the central imaging core laboratory on baseline NCCT, 24-hour NCCT, and the 96-hour scan (MRI and/or NCCT) and the scans obtained prior to DC, IPH evacuation, or CMO.
Time Frame: Baseline up to 96 hours (Day 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 38 | 20 | 19
mL
  Baseline | 22.41 (23.234) | 15.10 (16.366) | 17.52 (24.103)
  Change From Baseline at 96 Hours: number analyzed (Participants) | 34 | 19 | 15
  Change From Baseline at 96 Hours | 16.13 (20.872) | 25.87 (27.772) | 14.98 (10.459)
Statistical Analysis 1: Comparison: Placebo vs BIIB093 3 mg/Day vs BIIB093 5 mg/Day; Statistical analysis of combined BIIB093 vs placebo; Test type: Superiority; p = 0.6569, ANCOVA — P-value was analyzed by ANCOVA model with covariates: treatment, IRT stratification factors at randomization, baseline absolute edema volume based on central read, baseline GCS based on eCRF, and imaging modality at Hour 96 (MRI vs NCCT); LS Mean difference = 2.18, 95% CI 2-sided [-7.61 to 11.98]

8. Secondary Outcome: Time to All-Cause Death Through Day 90
Description: Time to all-cause death is defined as the time from randomization to the time of death and includes all-cause death along with neurological death.
Time Frame: Randomization up to Day 90
Population: mITT population included all randomized participants who received any study drug (BIIB093/placebo), had at least one final read per central review of contusion volume from NCCT or MRI scan acquired between 10 hours after study drug infusion initiation and Hour 96 visit or NSx or CMO, if earlier. 'Overall number of participants analyzed' signifies the number of participants who died from randomization up to Day 90.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | BIIB093 3 mg/Day | BIIB093 5 mg/Day
Number analyzed (Participants) | 3 | 0 | 1
days | NA [NA to NA] — Not estimable due to the small number of deaths. |  | NA [NA to NA] — Not estimable due to the small number of deaths.

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to last follow-up visit (approximately 1360 days)
Description: Safety analysis set included all randomized participants who had received any infusion of the study drug (BIIB093 or placebo).
Groups:
- BIIB093 3mg/Day: Participants were administered with BIIB093 up to 3 mg/day as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
- BIIB093 5mg/Day: Participants were administered with BIIB093 up to 5 mg/day as an IV bolus followed by a rapid IV infusion and a slow IV infusion for 4 days.
Arm/Group | Placebo | BIIB093 3mg/Day | BIIB093 5mg/Day
All-Cause Mortality (participants affected / at risk) | 4/44 | 0/23 | 2/19
Serious Adverse Events (participants affected / at risk) | 12/44 | 7/23 | 8/19
Other Adverse Events (participants affected / at risk) | 36/44 | 20/23 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | BIIB093 3mg/Day (N=23) | BIIB093 5mg/Day (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 4
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 0 | 3
Neurological decompensation (Nervous system disorders) | 1 | 0 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 0
Korsakoff's syndrome (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | BIIB093 3mg/Day (N=23) | BIIB093 5mg/Day (N=19)
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 2
Dilutional anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 1
Bradycardia (Cardiac disorders) | 5 | 4 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Anisocoria (Eye disorders) | 3 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 10 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 3
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5 | 1
Asthenia (General disorders) | 2 | 2 | 0
Generalised oedema (General disorders) | 1 | 0 | 1
Hypothermia (General disorders) | 4 | 0 | 0
Medical device site erosion (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 2 | 1
Pyrexia (General disorders) | 9 | 6 | 3
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 1
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 3 | 0
Covid-19 (Infections and infestations) | 2 | 0 | 1
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 9 | 3 | 3
Pneumonia aspiration (Infections and infestations) | 2 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 6 | 2 | 0
Electroencephalogram abnormal (Investigations) | 3 | 1 | 0
Fibrin d dimer increased (Investigations) | 4 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 5 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 2 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 7 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Anosmia (Nervous system disorders) | 3 | 2 | 0
Aphasia (Nervous system disorders) | 2 | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 2 | 0
Dementia with lewy bodies (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 2
Epilepsy (Nervous system disorders) | 3 | 2 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 7 | 4 | 2
Intracranial pressure increased (Nervous system disorders) | 5 | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Lateral medullary syndrome (Nervous system disorders) | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 3 | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Subdural hygroma (Nervous system disorders) | 1 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1
Agitation (Psychiatric disorders) | 6 | 1 | 3
Confusional state (Psychiatric disorders) | 2 | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1 | 3
Disorientation (Psychiatric disorders) | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 3 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0
Oliguria (Renal and urinary disorders) | 5 | 3 | 1
Polyuria (Renal and urinary disorders) | 5 | 1 | 0
Priapism (Reproductive system and breast disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Hypertension (Vascular disorders) | 9 | 6 | 4
Hypotension (Vascular disorders) | 6 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Early termination of trial due to strategic considerations, not for efficacy or safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03954041/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT03954041/SAP_001.pdf